CLINICAL TRIAL: NCT01122316
Title: Management of Diabetes With Metformin In Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Tamara Horwich, Tamara Horwich, MD, MS, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-06-086-02
Record Dates: First submitted 2010-05-12; First posted 2010-05-13 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure; Diabetes
Keywords: Heart Failure; Diabetes; Metformin
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 3. Metformin will be started at 500 mg PO BID and pending lab values may be titrated to 1000 mg PO BID at 1 month.

SUMMARY:
The Ahmanson-UCLA Cardiomyopathy Center is conducting a clinical research study that will assess the use of the medication metformin to improve quality of life, exercise capacity, and improved outcomes with patients that have both heart failure and diabetes.

If you participate in this study, you will receive the drug metformin for approximately 3 months. During the study you will undergo comprehensive testing which includes blood draws, an echocardiogram, and an magnetic resonance imaging (MRI)(if you do not have a pacemaker or defibrillator). You will also fill out a questionnaire and keep a blood glucose log.

You must be 18 years old to participate. The study drugs, study follow-up visits, and laboratory tests will be provided free of charge. Participants will be reimbursed up to $200 for their time and travel expenses.

DETAILED DESCRIPTION:
Heart failure (HF) affects 5 million individuals in the United States including over 10% of elderly persons >75 years. HF mortality is high, with approximately 20% 1-year risk of death (1). Diabetes (DM) is a common co-morbidity in patients with HF, present in approximately 25% of stable outpatients and 40% of hospitalized patients with HF (2). Diabetes in HF patients is associated with higher mortality (3,4). Hyperglycemia is independently associated with hospitalization for HF, longer length of stay during HF hospitalization, as well as higher in-hospital HF mortality (5-7). Furthermore, HF patients with more symptoms and worse functional status are more likely to have insulin resistance (8,9).

Despite the abundance of evidence linking diabetes, insulin resistance, and hyperglycemia to impaired functional status and worse outcomes in patients with HF, there is lack of data and guidelines on optimal strategies to manage diabetes in patients with chronic HF. In retrospective studies, many diabetes medications in HF have been associated with harm including insulin, thiazolidinediones, and sulfonylureas (10). The only anti-hyperglycemic medication that has been associated in retrospective studies with benefit in patients with HF and diabetes is metformin, which recently had its "black box warning" in HF lifted by the FDA, although most physicians are unaware of the change in labeling (10-12). Our analysis of data on 401 advanced, systolic HF patients with DM followed at the Ahmanson-UCLA Cardiomyopathy Center also found metformin therapy to be associated with improvement of left ventricular ejection fraction (LVEF) as well as decreased 1-year mortality (figure 1)(13).

Glycemic control in HF patients has not been prospectively studied; however, improved glycemic control has potential benefits in HF, including improvement of myocardial glucose utilization, decrease of potentially cardiotoxic free fatty acids, and reduced accumulation of myocardial collagen and advanced glycation end-products (14,15). Metformin therapy, compared to insulin and other antidiabetic medications, has potentially beneficial mechanisms of action in HF including insulin sensitization, improvement in lipid profiles, and more efficient myocardial metabolism (16,17). The purpose of this study is to gather pilot data for an anticipated comprehensive study DM management in HF, with the goal of NIH funding.

ELIGIBILITY:
Inclusion Criteria:

* Systolic HF of any etiology (left ventricular ejection fraction ≤ 40%)
* Previously-diagnosed, inadequately controlled DM (HbA1c≥7.5%)
* On any combination of anti-diabetic medications excluding metformin

Exclusion Criteria:

* Current metformin therapy
* Previous intolerance to metformin therapy
* Renal dysfunction (creatinine clearance < 60 ml/minute)
* History of lactic acidosis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Horwich, MD, MS, Principal Investigator — University of California, Los Angeles
Locations (1):
- Ahmanson-UCLA Cardiomyopathy Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Metformin at 500 mg PO BID and pending lab values may have been titrated to 1000 mg PO BID at 1 month.
Period: Overall Study
Arm/Group | Metformin
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Metformin
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Health-Related Quality of Life (HRQoL)
Description: HRQoL as assessed by the Minnesota Living With Heart Failure Questionnaire (MLHFQ)
  The MLHFQ is a self-administered questionnaire for patients with HF, comprising 21 items rated on six-point Likert scales, representing different degrees of impact of HF on HRQoL, from 0 (none) to 5 (very much). It provides a total score range 0-105. Lower scores indicate better health-related quality of life (HRQoL).
Time Frame: 3 months
Population: Analysis includes participants who completed intervention and final study assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metformin
Number analyzed (Participants) | 8
score on a scale
  Baseline | 56 (25)
  Three Months | 53 (35)

2. Secondary Outcome: Glycated Hemoglobin (HbA1c)
Description: The HbA1c test measures how much glucose is bound to hemoglobin in the red blood cells. The test shows the average level of glucose in blood for the past 3 months (the average lifespan of red blood cells). If glucose levels have been high over recent weeks, the hemoglobin A1c test will be higher.
Time Frame: 3 months
Population: Analysis includes participants who completed intervention and final study assessment
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Metformin
Number analyzed (Participants) | 8
percentage of glycated hemoglobin
  Baseline | 9.1 (2.3)
  Three Months | 8.9 (3.0)

3. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Obtained from Echocardiography
Time Frame: 3 months
Population: Analysis includes participants who completed intervention and final study assessment
Measure: Mean (Standard Deviation); unit: percent ejection fraction
Arm/Group | Metformin
Number analyzed (Participants) | 8
percent ejection fraction
  Baseline | 22 (11)
  Three Months | 28 (11)

4. Secondary Outcome: Creatinine Level as a Measure of Renal Function
Description: Serum creatinine
Time Frame: 3 months
Population: Analysis includes participants who completed intervention and final study assessment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin
Number analyzed (Participants) | 8
mg/dL
  Baseline | 1.04 (0.18)
  Three Months | 1.09 (0.2)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Metformin
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes